CLINICAL TRIAL: NCT05011370
Title: A Prospective Prevalence Study in Adolescent and Adult Patients Dependent on Parenteral Nutrition to Assess the Incidence of Intestinal Failure-Associated Liver Disease
Brief Title: Prevalence of Liver Disease in Patients Dependent on Parenteral Nutrition
Acronym: THRIVE-1
Status: Completed | Type: Observational
Sponsor: Protara Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: TARA-001-502
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Intestinal Failure-associated Liver Disease
Keywords: Intestinal failure-associated liver disease (IFALD); IFALD; Liver disease; Parenteral nutrition; Choline deficiency; Hepatic steatosis; Cholestasis; parenteral nutrition-associated liver disease
MeSH Terms: conditions — Liver Diseases; Hyperphagia; Choline Deficiency; Fatty Liver; Cholestasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center prospective cross-sectional observational study that will assess the prevalence of liver disease in patients dependent on parenteral nutrition (PN) for 4 or more days per week. Liver disease will be determined by the presence of choline deficiency, cholestasis (confirmed by elevated serum alkaline phosphatase (ALP) liver isoenzyme level), and steatosis (confirmed by magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF).

The objective of this study is to investigate the presence/prevalence of liver disease in patients dependent on PN (≥4 days a week).

DETAILED DESCRIPTION:
Eligible participants will provide blood samples at Visit 1 to determine choline deficiency, elevated serum ALP liver isoenzyme level and liver dysfunction, and complete one imaging study (MRI-PDFF) at Visit 1 to assess steatosis.

The purpose of this study is to understand and document critical epidemiological data related to choline deficiency and the incidence of liver disease in patients dependent on PN (≥ 4 days a week) and to better understand this patient population to help determine who might benefit from innovative treatments including IV Choline Chloride treatment.

ELIGIBILITY:
Inclusion Criteria:

* The participant and/or their parent/Legally Authorized Representative is willing and able to provide signed informed consent or assent as appropriate
* Male or female adults 18 to 80 years of age, or adolescents 12 to 17 years of age
* Patients dependent on parenteral nutrition (PN) that receive PN for an average ≥ 4 days a week for 10 weeks or longer prior to screening to meet nutritional, caloric, fluid, and/or electrolyte needs
* The Investigator expects no changes in the lipid, dextrose, amino acid, or vitamin regimen to be medically necessary during the participant's participation in the study
* Willingness of participant to maintain his/her current habitual oral diet and fluids regimen for the study duration

Exclusion Criteria:

* Participants taking steatogenic medications for ≥12 weeks in the past 12 months (e.g., amiodarone, tamoxifen, methotrexate, tetracycline, glucocorticoids, anabolic steroids, over the usual dose of estrogen for hormone replacement therapy, and valproate); those taking any medicine (e.g., metformin, thiazolidinediones, ursodeoxycholic acid, pentoxifylline, S-adenosyl-L-Methionine, and betaine) that could affect the measurement of IFALD within 12 weeks prior to study entry
* Participants taking potential hepatotoxic medications that in the judgement of the Investigator is causing hepatic abnormalities
* Participants with a cardiac pacemaker, intravascular stents, other metallic devices, and claustrophobia which are contraindicated to magnetic resonance imaging
* Participants who took choline supplements or choline-containing multivitamins within 14 days of screening
* History of major organ transplant (e.g., heart, kidney, liver, etc.)

For more information on eligibility criteria, please contact the sponsor.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll male and female adults and adolescent participants 12 years and older who are dependent on PN (≥ 4 days a week) in the primary care clinic setting.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with choline deficiency | Day 1
  Choline deficiency is defined as plasma-free choline concentration less than 7 nmol/mL.
Percentage of patients with choline deficiency, elevated serum ALP liver isoenzyme level and MRI-PDFF ≥8% | Day 1
  Choline deficiency is defined as plasma-free choline concentration less than 7 nmol/mL. Elevated serum ALP liver isoenzyme level is defined as >1.5x upper limit of normal. MRI-PDFF ≥8 %

SECONDARY OUTCOMES:
Percentage of patients with MRI-PDFF ≥8% | Day 1
  Assessment of liver tests all patients and patients with choline deficiency. Choline deficiency is defined as plasma-free choline concentration less than 7 nmol/mL;
Percentage of patients with elevated serum ALP liver isoenzyme level (defined as ≥ 1.5x upper limit of normal) | Day 1
  Assessment of liver tests all patients and patients with choline deficiency. Choline deficiency is defined as plasma-free choline concentration less than 7 nmol/mL;
Percentage of patients with abnormal liver tests including serum direct bilirubin, AST, ALT and GGT | Day 1
  Assessment of liver tests all patients and patients with choline deficiency. Choline deficiency is defined as plasma-free choline concentration less than 7 nmol/mL; AST = aspartate aminotransferase; ALT = alanine transaminase; GGT = gamma-glutamyl transferase.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Operations Officer, Study Director — Protara Therapeutics
Locations (15):
- United States (10):
  - Ronald Reagan Medical Center of UCLA, Los Angeles, California
  - IHS Health, Kissimmee, Florida
  - The University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's, Seattle, Washington
- Rigshospitalet, Copenhagen, Denmark
- Center for Chronic Intestinal Failure, St. Orsola Hospital Dept of Medical and Surgical Sciences, University of Bologna, Bologna, Italy
- United Kingdom (3):
  - St. Mark's Hospital, Harrow, England
  - University College London Hospitals, London, England
  - Northern Care Alliance NHS Foundation, Salford, England

IPD SHARING:
Plan to Share IPD: No